CLINICAL TRIAL: NCT02350036
Title: Maternal Serum Placental Protein 13 Serum Endoglin and Uterine Doppler Indeces as Predictors of Pre-eclampsia and Relation to Maternal and Neonatal Outcome
Brief Title: Placental Protein 13 Serum Endoglin and Uterine Doppler Indeces as Predictors of Pre-eclampsia
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Other Study IDs: 125
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; placental protein 13; Uterine artery doppler
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- preeclmapsia: women developed preeclampsia. ultrasound monitoring and uterine artery Doppler
  Interventions: Other: ultrasound monitoring
- control: women with normal blood pressure all through pregnancy. ultrasound monitoring and uterine artery Doppler
  Interventions: Other: ultrasound monitoring

INTERVENTIONS:
Other: ultrasound monitoring — Uterine artery Doppler assessment

SUMMARY:
50 pregnant females were divided in two groups, twenty five as a control group and twenty five as high risk group; they were subjected to uterine artery Doppler, measurement of maternal serum and detection of (MTHFR) gene polymorphisms in first trimester at 11 to 14 weeks of gestation, all pregnancies were followed until 40 weeks for development of pre-eclampsia

DETAILED DESCRIPTION:
50 pregnant females were divided in two groups, twenty five as a control group and twenty five as high risk group; they were subjected to uterine artery Doppler, measurement of maternal serum (pp-13) and detection of (MTHFR) gene polymorphisms in first trimester at 11 to 14 weeks of gestation, all pregnancies were followed until 40 weeks for development of pre-eclampsia

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at 11 to 14 weeks of gestation

Exclusion Criteria:

* fetal anomalies other medical diseases as diabetes mellitus, renal or liver diseases

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women at 11 to 14 weeks of gestation
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
development of preeclampsia | 40 weeks pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt